CLINICAL TRIAL: NCT03131336
Title: A Controlled, Randomized, Multi-centre, Double Blind, Phase II Study to Evaluate Efficacy and Safety of Topical PeproStat in Intraoperative Surgical Haemostasis
Brief Title: PeproStat as a Topical Agent Used to Stop Bleeding in Patients Undergoing Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Haemostatix Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HX-02-PEP
Record Dates: First submitted 2017-03-27; First posted 2017-04-27 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Bleeding
MeSH Terms: conditions — Hemorrhage | interventions — Sodium Chloride; Gelatin Sponge, Absorbable; Fibrin Foam

STUDY DESIGN:
Intervention Model Description: Prospective, interventional, randomized, controlled, double-blind, parallel group
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PeproStat (Experimental): PeproStat 2.5mg/mL soaked into haemostatic gelatin sponge, applied to a target bleeding site
  Interventions: Drug: PeproStat
- Saline (Placebo Comparator): Saline soaked into haemostatic gelatin sponge, applied to a target bleeding site
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: PeproStat — solution for local application
  Other Names: PeproStat 2.5 mg/mL, soaked into Spongostan
  Arms: PeproStat
Drug: Saline — solution for local application
  Other Names: Absorbable gelatin sponge (Spongostan) soaked with saline
  Arms: Saline

SUMMARY:
The purpose of this study is to test the effectiveness and safety of a new peptide-based coagulant, PeproStat. The study drug will be applied to patients undergoing liver/soft tissue surgery, vascular surgery or spine surgery. The speed of action of the new coagulant, that is applied with a gelatin sponge, will be compared to the same sponge but with saline (a commonly used standard of care).

DETAILED DESCRIPTION:
PeproStat is a new class of topical haemostatic agent composed of recombinant human albumin (rHA) conjugated with fibrinogen-binding peptides. The conjugate polymerises fibrinogen into a fibrin-like clot without the need for thrombin.

PeproStat is formulated in a liquid, and is soaked into a haemostatic gelatin sponge in the operating theatre, and applied directly to the site of bleeding. The gelatin sponge (Spongostan ) is an approved "passive" haemostat i.e., PeproStat is an adjunct to a passive haemostat.

The study is designed in a 2:1 randomization (verum:placebo) to investigate the efficacy in terms of Time to hemostasis, mean (mTTH) at the primary target bleed site (TBS), measured in minutes (min) from the start of treatment application (TxStart) at the TBS to the achievement of hemostasis at that site or to the end of the 10-minute assessment period if hemostasis has not yet been achieved.

ELIGIBILITY:
Inclusion Criteria: At screening and baseline:

1. Subject is undergoing a planned open liver/soft tissue surgery, vascular surgery or spine surgery.
2. Subjects are able and willing to provide written informed consent to participate in this study.
3. Adult males and females ≥18 years of age at screening.
4. Willing and able to comply with all protocol requirements including follow-up assessments.
5. Male subjects must be willing and able to use adequate contraception from enrollment through to the 30 day follow-up visit.
6. Women of childbearing potential (WCBP)C have to use highly effective methods of contraception from enrollment through to the 30 day follow-up visit.

   Intraoperative:
7. The subject presents an identified target bleeding site with mild or moderate bleeding, which conventional surgical techniques are insufficient to control or are inappropriate and would otherwise be a candidate for standard haemostats.
8. The subject presents no intraoperative complications, other than bleeding, that may interfere with study assessments as judged by the Investigator.
9. The subject presents no contaminated areas of the body, signs of infection or abscess development.
10. Total target bleeding site surface area of ≤ 70 cm2, defined within one or two TBSs.

Exclusion Criteria:

1. Subject is undergoing emergency surgical procedure.
2. Use of study treatment and sponge in

   * Closure of skin incisions as the sponge may interfere with the healing of skin edges.
   * Intravascular compartments because of the risk of embolization following sponge application.
3. Recipient of an organ transplant.
4. Haematologic, biochemistry and coagulation panel thresholds at screening:

   * Haemoglobin ≤ 9.0 g/dL.
   * Platelet count ≤100,000/mm3 (≤ 100 x 109/L).
   * International Normalized Ratio (INR) > 2.0 or activated Partial Thromboplastin Time (aPTT) ratio > 2.0.
   * Fibrinogen level < 1.5 g/L.
   * Aspartate Aminotransferase (AST) or Alanine aminotransferase (ALT) ≥ 3 times the upper limit normal range, except for subjects undergoing liver resection surgery where there is no upper limit for these analytes due to the nature of their disease.
5. Severe renal failure.
6. Any other disease or condition that may affect normal blood clotting, for example thrombocytopenia, as judged by the Investigator.
7. A known history of anaphylaxis or allergic reaction to human albumin, PEGylated proteins, yeast or moulds, porcine products or other components in the study medication or sponge.
8. Participation in another investigational drug or device research study within 30 days before and after enrolment in the current study.
9. Current known or suspected alcohol and/or drug abuse or dependence at the time of screening.
10. Any concurrent medical, surgical, or psychiatric condition that may, in the Investigator's opinion, affect the subject's willingness or ability to meet all study requirements during the study duration.
11. Known HIV, Hepatitis B virus or Hepatitis C Virus infection.
12. During the surgery, subject presents severe bleeding where use of a topical haemostat would be inappropriate.
13. Anti-platelets/oral anticoagulants treatment:

    1. Soft tissue/liver and neurosurgery: Subject is taking anti-platelet agents or oral anticoagulants within 7 days of surgery
    2. Vascular surgery: Subject is taking dual anti-platelet treatment or oral anticoagulants within 7 days of surgery. One anti-platelet agent is allowed perioperatively.
14. Heparin treatment:

    c. Soft tissue/liver and neurosurgery only: Subject is receiving therapeutic doses of heparin perioperatively. Only prophylactic Low Molecular Weight Heparin is allowed.
15. Pregnant or breast-feeding subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2017-08-23 (Actual); Study Completion 2017-10-11 (Actual)

PRIMARY OUTCOMES:
The difference in time to hemostasis in minutes when using verum vs placebo | 10 minutes after application
  Efficacy in terms of Time to hemostasis, mean (mTTH) at the primary target bleed site (TBS),measured in minutes from the start of treatment application (TxStart) at the TBS to the achievement of haemostasis at that site or to the end of the 10-minute assessment period if haemostasis has not yet been achieved.

SECONDARY OUTCOMES:
Percentage of subjects achieving hemostasis at 1 min haemostasis in adult subjects undergoing open liver/soft tissue, vascular and spine surgery using descriptive statistics | 1 minute after start of treatment
  Percentage of subjects achieving haemostasis within 1 minute from application of treatment
Percentage of subjects achieving hemostasis at 2 min haemostasis in adult subjects undergoing open liver/soft tissue, vascular and spine surgery using descriptive statistics | 2 minutes after start of treatment
  Percentage of subjects achieving haemostasis within 2 minutes from application of treatment
Percentage of subjects achieving hemostasis at 3 min haemostasis in adult subjects undergoing open liver/soft tissue, vascular and spine surgery using descriptive statistics | 3 minutes after start of treatment
  Percentage of subjects achieving haemostasis within 3 minutes from application of treatment
Percentage of subjects achieving hemostasis at 5 min haemostasis in adult subjects undergoing open liver/soft tissue, vascular and spine surgery using descriptive statistics | 5 minutes after start of treatment
  Percentage of subjects achieving haemostasis within 5 minutes from application of treatment
Percentage of subjects achieving hemostasis at 7 min haemostasis in adult subjects undergoing open liver/soft tissue, vascular and spine surgery using descriptive statistics | 7 minutes after start of treatment
  Percentage of subjects achieving haemostasis within 7 minutes from application of treatment
Percentage of subjects achieving hemostasis at 10 min haemostasis in adult subjects undergoing open liver/soft tissue, vascular and spine surgery using descriptive statistics | 10 minutes after start of treatment
  Percentage of subjects achieving haemostasis within 10 minutes from application of treatment
Median time to hemostasis in minutes from TxStart to the achievement of hemostasis or to the end of the 10-minute assessment period if hemostasis has not yet been achieved | 10 minutes after start of treatment
  Median time for haemostasis to be achieved
Number/rate of subjects who do not achieve hemostasis within 10 min | 10 minutes after start of treatment
  Number/rate of subjects who do not achieve hemostasis within 10 min
Number of sponges applied at Target Bleeding Site (TBS) | Counted on Day of surgery
  Number of sponges used at TBS, 1 or 2
Dose of PeproStat determined by number and size (if cut to size) of PeproStat soaked sponges applied at TBS | Measured on day of surgery
  Dose of PeproStat determined by number and size (if cut to size) of PeproStat soaked sponges applied at TBS
Number/rate of treatment failures | 10 minutes after start of treatment
  Number of participants not achieving haemostasis within 10 minutes at primary, secondary or both TBS's
Use of alternative haemostatic agents at the TBS | Documented on the day of surgery
  Number of participants requiring use of other haemostats at the TBS
Investigator assessment of efficacy to obtain haemostasis | Documented on the day of surgery
  Investigator's assessment of the efficacy of the treatment with a score of 1-5, where 5 is very effective
Investigator assessment ease of use of study treatment | Documented on the day of surgery
  Investigator assessment ease of use of study treatment with a score of 1-5, where 5 is very effective
Adverse Events | Measured from the point of consent to Day 30
  Number of Adverse Events (AEs) including adverse events of special interest: Bleeding at the TBS after 10-minute assessment period during or after surgery (if re-operation is required) and transfusion requirement
Heparin usage | Measured from the point of consent to Day 30
  Number of participants with Heparin usage
Antiplatelet usage | Measured from the point of consent to Day 30
  Number of participants with Antiplatelet usage
Laboratory safety parameters | Measured at Day 5
  Changes in Laboratory safety parameters at day 5 vs. screening
Laboratory safety parameters | Measured at screening, Day 30
  Laboratory safety parameters at day 30 vs. screening
Immunogenicity testing | Measured at screening and Day 30
  Immunogenicity testing
Vital signs | Measured before surgery vs. screening
  Changes in vital signs
Vital signs | Measured during surgery (before treatment) vs. screening
  Changes in vital signs
Vital signs | Measured during surgery (15 minutes after treatment) vs. screening
  Changes in vital signs
Vital signs | Measured at 4 hours after surgery vs. screening
  Changes in vital signs
Vital signs | Measured at 8 hours after surgery vs. screening
  Changes in vital signs
Vital signs | Measured at 16 hours after surgery vs. screening
  Changes in vital signs
12-lead electrocardiogram | measured at Day 5
  Abnormalities in 12-lead electrocardiogram
12-lead electrocardiogram | measured at Day 30 (if medically indicated)
  Abnormalities in 12-lead electrocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Paul Hayes, Principal Investigator — Addenbrookes NHS Trust
Locations (5):
- University Clinical Hospital, Bolnicka 25, Sarajevo, Bosnia and Herzegovina
- University Clinical Hospital Centre "Sestre Milosrdnice", Vinogradska cesta 29, Zagreb, Croatia
- Klinika Neurochirurgii Gdanskie Centrum Kliniczne, ul. Dębinki 7, Gdansk, Poland
- Clinical centre of Serbia, Clinic for vascular and endovascular surgery, Koste Todorovica Street 8, Belgrade, Serbia
- Addenbrookes Hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No